CLINICAL TRIAL: NCT00343603
Title: Tracking Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0309019; 2R44EY013036 (NIH)
Record Dates: First submitted 2006-06-19; First posted 2006-06-23 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2011-07

CONDITIONS: Macular Degeneration; Glaucoma; Diabetic Retinopathy; Choroidal Disease
Keywords: maculopathy
MeSH Terms: conditions — Macular Degeneration; Glaucoma; Diabetic Retinopathy; Choroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to evaluate an investigational system that may allow doctors to show images of the different parts inside the eye that show greater detail than current equipment can produce.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate an investigational system that may allow doctors to make images of the parts inside the eye that show greater detail than current equipment can produce.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (this includes women of child-bearing potential) who are familiar with vision experiments and ophthalmic equipment, all over 18 years.
* Subjects will have a retinal screening if they are over 50 years old or have a known risk factor for eye disease, such as family history of age related macular degeneration or cardiovascular disease.
* Patients with retinal and choroidal disease: age related maculopathy or age related macular degeneration, diabetic retinopathy, glaucoma.

Exclusion Criteria:

* Over 85 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject can range between 18 to 85 years old. They can be healthy or diseased. Recruiting males and females.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gadi Wollstein, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided